CLINICAL TRIAL: NCT04885842
Title: Evaluation of the Efficacy of Injection Platelet-rich Fibrin(I-PRF) in Accelerate Alignment and Leveling in an Adult Sample
Brief Title: Efficacy of Injection Platelet-rich Fibrin(I-PRF) in Accelerate Alignment and Leveling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TishreenU
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-03

CONDITIONS: Orthodontic Pathological Resorption of External Root
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical study ,two parallel groups design. The research sample consisted of 18 patients (11 famales,7 males)Patients were randomly assigned to 2 groups using the sample randomization principle. Each group included 8 patient (9 control group applying brackets only)(9 group injection I-PRF with brackets).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): injection I-PRF with brackets
  Interventions: Other: injection I-PRF
- Control Group (No Intervention): applying brackets only

INTERVENTIONS:
Other: injection I-PRF — injection I-PRF with brackets
  Other Names: control Group
  Arms: Study Group

SUMMARY:
the aim of this study is to evaluate the effectiveness of injection I-PRF to accelerate alignment and leveling of the upper anterior teeth and reduce the time required for treatment.

DETAILED DESCRIPTION:
What remains the most important and common question for adult patients who want to undergo orthodontic treatment is how long the treatment will take, as the period of orthodontic treatment may take between 18 and 24 months in some cases of malocclusion ,and this may cause discomfort for the patient and reduce cooperation during treatment in addition to the aesthetic problems associated with presence of bracket.

the possibility of an increase of Enamel mineral dissolution and spread of dental caries ,gingival problems and this is due to the increase of the duration of orthodontic treatment.

Orthodontic treatment begins with the leveling and alignment stage and constitutes an important part of the treatment stages, during which the teeth(incisal edges, cusps posterior teeth) are placed on one level and to achieve perfect points of contact between the teeth In some cases of malocclusion especially severe ones, this stage may take about 8 months therefore , the interest of orthodontics has increased in finding new methods and techniques in order to accelerate treatment, Various methods and techniques have been used to accelerate orthodontic treatment Which includes :biomaterial injection, surgical and physical methods. Yet, despite the effectiveness of some of these methods in accelerating dental movement ,each of its disadvantages and side effects on the patient therefore, attention must be paid to anther effective safe and simple non-traumatic method hence the idea of using platelet rich fibrin came.

Platelet rich fibrin is a therapeutic approach and it is a new generation of platelet concentrates Which was introduced to the field of dentistry by choukroun in 2001 who developed this treatment technique.

Platelet rich fibrin injection technology (I-PRF), which is obtained in liquid form for injection has been developed through the concept of reduced speed centrifugation .

PRF is a biomaterial .Autologus is taken from a person's own blood.Unlike PRP, no external bioactive are added to active platelet. Rather, the blood sample remains normal. The importance and therapeutic benefits of platelet-rich fibrin come through the presence of key and other common elements that collectively contribute to the healing processes and regeneration of the soft and bone tissues represented by the presence of fibrin in the form of a matrix with large and significant numbers of leukocytes, cytokines, platelets, in addition to the participation of growth factors which play an important role in the processes of healing.

Platelet rich fibrin is a simple, easy to apply and economical technique that does not require adding any substances to the blood sample as an anticoagulant.

To date, there are no studies on the role that platelet rich fibrin injection can play in accelerating aligning and leveling the upper anterior teeth and reducing the time required for treatments Therefore the aim of study is to verify the effectiveness of injection I-PRF to accelerate alignment and leveling of the upper anterior teeth and reduce the time required for treatment

ELIGIBILITY:
Inclusion Criteria:

The Clinical Diagnosis the age of patients ranges between 16-24 years, medium crowding between 3-6 mm in the area of the upper anterior teeth according to Little irregularity index 20,class1 according angel classification,

Exclusion Criteria:

the presence of any systemic disease that affects the orthodontic movement Diabetes , a patient undergoing previous orthodontic treatment, a patient who takes medicines Cortisone,NSAIDs the affect dental movement . and the presence of bleeding disorders Disturbance in the number of platelets.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2019-09-14 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
alignment and leveling Improvement Percentage(ALIP): | 6 Month
  Determining the percentage of improvement in alignment and leveling by calculating the value of the change in the Little index in one of the studied time periods (T1) or (T2) or (T3) which is calculated by subtracting the value of the Little index at the studied period of time from the value of the Little index at (T0) When the primary wire is inserted, the value of the little index at (T0) is multiplied by 100 Through the following

SECONDARY OUTCOMES:
Overall Alignment and Leveling Time | 6 Month
  the overall time required to complete the leveling and alignment was calculated by calculating the number of days between (To) and (T3).

CONTACTS AND LOCATIONS:
Locations (1):
- Tishreen University, Latakia, Syria

REFERENCES:
- [Result] The gliding path of the mandible along the skull. Ferdinand Graf Spee (1855-1937), prosector at the Anatomy Institute of Kiel. J Am Dent Assoc. 1980 May;100(5):670-5. No abstract available. PMID 6988491
- [Result] Baldridge DW. Leveling the curve of Spee: its effect on mandibular arch length. JPO J Pract Orthod. 1969 Jan;3(1):26-41. No abstract available. PMID 5250875
- See also: Introducing Choukroun's platelet rich fibrin (PRF) to the reconstructive surgery milieu. J Implant Adv Clin Dent 2009;1:21-30 — http://www.academia.edu/15581747/